CLINICAL TRIAL: NCT06433830
Title: A Single-arm, Phase II Trial of Hetrombopag for the Treatment of Concurrent Chemoradiotherapy-induced Thrombocytopenia in Patients With Advanced Solid Tumors
Brief Title: Hetrombopag for the Thrombocytopenia Induced by Concurrent Chemoradiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20220125-10
Record Dates: First submitted 2024-04-29; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Thrombocytopenia; Radiotherapy Side Effect
Keywords: hetrombopag; thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia; Radiation Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hetrombopag (Experimental): patients receive oral hetrombopag at an initial dose of 7.5 mg QD
  Interventions: Drug: Hetrombopag Olamine

INTERVENTIONS:
Drug: Hetrombopag Olamine — The administration of hetrombopag as a monotherapy and at an initial dose of 7.5 mg QD.The dose adjusted based on platelet count.
  Other Names: thrombopoietin receptor agonist

SUMMARY:
Thrombocytopenia represents one of the main toxicities of concurrent chemoradiotherapy, which may necessitate chemotherapy dose reductions, dose delays, or discontinuation, and even compromise survival. Hetrombopag, a thrombopoietin receptor agonist, has shown efficacy and safety in patients with chemotherapy-induced thrombocytopenia. However, the efficacy of hetrombopag in patients who received concurrent chemoradiotherapy is not clear yet. This study aimed to evaluate the efficacy and safety of hetrombopag in this patient population.

DETAILED DESCRIPTION:
Antitumor related therapy is one of the common causes of thrombocytopenia. Chemotherapy regimens based on drugs such as gemcitabine, platinum, anthracycline, and paclitaxel are high-risk options for thrombocytopenia. The degree of thrombocytopenia caused by external radiation therapy mainly depends on the irradiation dose, irradiation site, irradiation field size, and irradiation duration. The synchronous radiotherapy and chemotherapy regimen for head and neck tumors, esophageal cancer, rectal cancer, and other cancers often involves platinum drugs, and the irradiation site often involves flat and irregular bones. Therefore, the incidence of thrombocytopenia in patients during the treatment process is higher than that of chemotherapy or radiotherapy alone. In a phase III clinical study on the combination of carboplatin and paclitaxel in the treatment of esophageal cancer, the incidence of thrombocytopenia was as high as 54%. Once thrombocytopenia occurs, it may lead to a decrease in chemotherapy drug dosage, delay, and cessation of radiotherapy and chemotherapy, and may require platelet infusion. In follow-up studies of various cancer patients, it has been found that reducing the dosage of chemotherapy drugs or delaying the chemotherapy cycle will reduce treatment efficacy and lead to poor prognosis, including shortened disease-free survival (DFS) and overall survival (OS) time.

TPO-RA drugs are currently approved for indications in the fields of chronic primary immune thrombocytopenia (ITP), severe aplastic anemia (SAA), and chronic liver disease (CLD). There are also relevant data reports in the CIT field. A phase II clinical study using romiplostim for the treatment of CIT enrolled a total of 60 patients. After treatment with romiplostim, 85% of patients returned to normal platelet count within 3 weeks and resumed chemotherapy. In the subsequent prescribed chemotherapy cycle, only 6.8% of patients experienced a relapse due to another round of chemotherapy. The occurrence of CIT leads to a decrease or delay in chemotherapy dose; In another randomized placebo-controlled phase II study using eltrombopag for the prevention of solid tumor CIT, patients received gemcitabine monotherapy or gemcitabine combined with cisplatin/carboplatin regimen chemotherapy, and treated with eltrombopag or placebo 100mg before and 5 days after chemotherapy. In the 1-6 chemotherapy cycles, the average platelet count on the day before chemotherapy in the eltrombopag group was numerically higher than that in the placebo group, but did not reach statistically significant differences. The incidence of grade 3/4 thrombocytopenia in the eltrombopag group was lower than that in the placebo group. Among patients in the combination chemotherapy group, the average time required for eltrombopag group to recover from the lowest platelet count to normal was 8 days. The placebo group, on the other hand, requires 15 days, and the incidence of delayed/reduced chemotherapy dose or dose loss due to thrombocytopenia is lower in patients in the eltrombopag group, Therefore, in gemcitabine based chemotherapy, treatment with eltrombopag can shorten the time for platelet minimum recovery and reduce the delayed/reduced chemotherapy dose caused by thrombocytopenia. However, there is still a lack of stronger evidence-based medicine for the application of TPO-RA drugs in CIT, and there is no relevant data in the field of concurrent chemoradiotherapy induced thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, regardless of gender;
* Malignant tumor patients diagnosed through pathological or cytological examination, regardless of cancer type, may experience thrombocytopenia during radical synchronous radiotherapy and chemotherapy treatment;
* Platelet count of patients ≤ 75 × 10^9/L on the day or 3 days prior to enrollment;
* Expected survival time ≥ 12 weeks;
* ECOG PS score for physical condition: 0-2 points;
* The laboratory inspection indicators meet the following requirements:

  1. Renal function: Cr ≤ ULN (upper limit of normal value) x 1.5, endogenous creatinine clearance rate (Ccr) ≥ 55 ml/min;
  2. Liver function: Total bilirubin ≤ ULN × 1.5; ALT and AST ≤ ULN × 3; (If it is intrahepatic cholangiocarcinoma or liver metastasis, total bilirubin should not exceed 3 times the normal upper limit, and transaminase should not exceed 5 times the normal upper limit);
* Women of childbearing age agree to use contraception during the study period and within 6 months after the end of the study; And not a lactating patient; Male patients who agree to contraception during the study period and within 6 months after the end of the study;
* Those who have not participated in clinical trials of other drugs within the 4 weeks prior to enrollment;
* It is expected that those with good compliance will be able to follow up on therapeutic effects and adverse reactions according to the protocol requirements;
* No serious complications such as active gastrointestinal bleeding, perforation, jaundice, gastrointestinal disorders Obstruction, non cancerous fever>38 °C;
* The subjects are able to understand the situation of this study and voluntarily sign an informed consent form.

Exclusion Criteria:

* Screening for thrombocytopenia caused by non tumor treatment within the first 6 months, including but not limited to liver cirrhosis, splenic hyper function, infection, and bleeding;
* Suffering from other hematopoietic system diseases besides thrombocytopenia caused by concurrent radiotherapy and chemotherapy for malignant tumors, including leukemia, primary immune thrombocytopenia, myeloproliferative diseases, multiple myeloma, and myelodysplastic syndrome;
* Combined bone marrow invasion or bone marrow metastasis;
* After treatment with infusion of red blood cells or erythropoietin (EPO), hemoglobin remains below 50g/L, or after treatment with granulocyte colony-stimulating factor (G-CSF), the absolute value of neutrophils remains below 1.0 × 10^9/L;
* Have received pelvic and spinal radiation therapy, as well as bone field radiation, within the three months prior to screening;
* History of arterial or venous thrombosis within the first 6 months of screening;
* Clinical manifestations of severe bleeding (such as gastrointestinal bleeding) within the first two weeks of screening;
* Received platelet transfusion within 2 days prior to enrollment;
* Screening for patients with severe cardiovascular diseases (such as NYHA heart function score III-IV), known arrhythmias that increase the risk of thromboembolism, such as atrial fibrillation, coronary stent implantation, angioplasty, and coronary artery bypass grafting within the first 6 months;
* Received treatment with recombinant human thrombopoietin (rhTPO), recombinant human interleukin-11 (rhIL-11), or thrombopoietin receptor agonists (such as eltrombopag, avatrombopag) within 14 days prior to screening;
* Patients who are known or expected to be allergic or intolerant to the active ingredients or excipients of hetrombopag tablets (excipients include cellulose lactose, low substituted hydroxypropyl cellulose, magnesium stearate, and film coated premixes);
* Breastfeeding women;
* Vulnerable groups, including individuals with mental illness, cognitive impairment, critically ill patients, minors, pregnant women, etc;
* The researcher believes that the participants are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with PLT ≥100×10^9/L | From admission to discharge, up to 6 weeks
  The response rate is defined as the proportion of patients who receive treatment with hetrombopag until PLT≥100×10^9/L

SECONDARY OUTCOMES:
The median time of PLT ≥100×10^9/L | From admission to discharge, up to 6 weeks
  Use Kaplan Meier method to estimate median platelet recovery time.
Incidence of delayed radiotherapy cycles due to thrombocytopenia | From admission to discharge, up to 6 weeks
  The number of events in which radiotherapy and chemotherapy were suspended due to thrombocytopenia, as determined by researchers
Number and percentage of patients receiving platelets transfusion for thrombocytopenia | From admission to discharge, up to 6 weeks
  Researchers determine the number of platelet transfusion events caused by thrombocytopenia
Incidence of serious adverse events according to CTCAE 5.0 criteria | From admission to the end of the study, up to 9 weeks
  Record the name and frequency of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Sun, Principal Investigator — Sir Run Run Shaw Hospital; Weiwen Zhou, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China